CLINICAL TRIAL: NCT06588114
Title: Antistress Ball Applied to Hemodialysis Patients, Valsalva Maneuver and Pain Due to Arteriovenous Fistula Cannulation of Skin Cooling Device and the Effect of Fear of Pain: a Randomized Controlled Trial
Brief Title: Arteriovenous Fistula Cannulation Pain and Skin Cooling Device
Acronym: HD patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karadeniz Technical University (Other)
Collaborators: Gümüşhane Universıty (Other)
Responsible Party: Principal Investigator, AYNUR CİN, Principal Investigator, Gümüşhane Universıty
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: E-95674917-108.99-248196
Record Dates: First submitted 2024-09-02; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Chronic Kidney Disease on Hemodialysis
Keywords: Hemodialysis; Arteriovenous fistula; Valsalva; Antistress ball
MeSH Terms: conditions — Arteriovenous Fistula

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- experimental group (skin cooler device) (Experimental): Hemodialysis patients in this group will be provided with skin temperature reduction by the researcher with a skin cooling device for 10 minutes before the arteriovenous fistula attempt is made.
  Interventions: Other: Skin cooling
- experimental group (Antistress Ball Group) (Experimental): Hemodialysis patients in this group will be asked to look away by giving an antistress ball to the non-arteriovenous fistula hand and squeezing and then loosening the ball during the arteriovenous fistula intervention.
  Interventions: Other: Antistress Ball
- experimental group (Valsalva Maneuver Group) (Experimental): The Valsalva maneuver is a breathing method that can slow down a heart with a very fast pulse rate. In this maneuver, the individual breathes strongly through his mouth while his nose is tightly closed, and while holding his breath, a strong tension occurs. This maneuver allows the heart to react and return to a normal rhythm. Hemodialysis patients in this group will perform the valsalva maneuver taught to them by the researcher during arteriovenous intervention.
  Interventions: Other: The Valsalva maneuver
- control group (No Intervention): Hemodialysis patients aged 18 years and older who have arteriovenous fistula and have been on hemodialysis for more than three months will be included in the control group. No intervention will be made to the control group. Patients in this group will receive routine check-ups and hemodialysis treatments.

INTERVENTIONS:
Other: Antistress Ball — Hemodialysis patients will be asked to look away by giving an antistress ball to the non-arteriovenous fistula hand and squeezing and then loosening the ball during the arteriovenous fistula intervention
  Arms: experimental group (Antistress Ball Group)
Other: The Valsalva maneuver — The Valsalva maneuver is a breathing method that can slow down a heart with a very fast pulse rate. In this maneuver, the individual breathes strongly through his mouth while his nose is tightly closed, and while holding his breath, a strong tension occurs. This maneuver allows the heart to react and return to a normal rhythm.
  Arms: experimental group (Valsalva Maneuver Group)
Other: Skin cooling — Hemodialysis patients will be provided with lowering of skin temperature with a skin cooling device by the researcher for 10 minutes before arteriovenous fistula intervention is made to hemodialysis patients
  Arms: experimental group (skin cooler device)

SUMMARY:
To determine the effect of the antistress ball, valsalva maneuver and skin cooling device, which are one of the nonpharmacological methods applied to hemodialysis patients, on the level of pain and fear of pain due to arteriovenous fistula cannulation.

DETAILED DESCRIPTION:
Patients with chronic renal failure who are being treated with hemodialysis experience pain during invasive intervention with arteriovenous fistula. This condition negatively affects hemodialysis patients and leads to a decrease in their quality of life. In order to reduce the pain and fear experienced during arteriovenous fistula intervention, it is recommended to use pharmacological methods as well as nonpharmacological methods. Antistress ball, which is one of the nonpharmacological methods, reduces pain during arteriovenous fistula intervention by causing distraction in hemodialysis patients, but its effect on fear of pain is not yet known. Of the other nonpharmacological methods, the valsalva maneuver reduces pain during vascular intervention, but the pain and fear of pain during arteriovenous fistula intervention have not yet been investigated. In the same way, the effects of skin cooling device on pain and fear of pain during arteriovenous fistula intervention are unknown. The aim of this randomized controlled trial is to; to determine the effect of the antistress ball, valsalva maneuver and skin cooling device, which are one of the nonpharmacological methods applied to hemodialysis patients, on the level of pain and fear of pain due to arteriovenous fistula cannulation. This study will be conducted in an experimental type and 60 patients receiving hemodialysis treatment at X State Hospital hemodialysis unit will form the sample of the study. All patients in the experimental group will be given nonpharmacological applications (antistress ball, valsalva maneuver and skin cooling application) for 8 weeks, three times a week. The control group will not be given any intervention and will receive routine treatment. The 'Pain Catastrophization Scale' will be applied to the experimental and control groups before, in the middle and after the research. The 'Visual Analog Pain Scale" will be used to determine the pain severity of hemodialysis patients before and after arteriovenous fistula intervention.

ELIGIBILITY:
Inclusion Criteria:

* be 18 years of age or older
* Volunteering to participate in the study
* Being a hemodialysis patient and being on hemodialysis for more than three months
* Having an arteriovenous fistula that has been used for more than a month
* To be hemodialyzed three times a week
* To be literate
* Absence of communication barrier
* Not having any psychiatric diagnosis
* Not having cognitive impairment

Exclusion Criteria:

* being under the age of 18
* It takes less than a month for the arteriovenous fistula to be newly opened
* Having a different type of vascular interference from arteriovenous fistula
* Having phlebitis, scar tissue, dermatitis, an incision or infection at the site of arteriovenous interference
* Hemodialysis of the patient more or less than three times a week
* Having any disease that may affect the perception of pain
* Illiteracy
* Having a psychiatric diagnosis
* Having any discomfort in the hand and arm that allows squeezing the antistress ball
* There is a communication barrier
* Having a cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2024-11-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Experimental group (skin cooling) The Pain Catastrophization Scale | 4 week
  This scale, developed by Sullivan et al. (1995), serves to measure the exaggerated negative mental reaction of individuals to an existing or predicted painful experience; to what extent they catastrophize the pain in the form of self-information . The reliability and validity of the Turkish version of the scale, which was shown by Uğurlu and others (2017), consists of 13 items. Each item is scored as none at all=0, mild degree=1, moderate degree=2, major degree=3 and always=4. A high total score indicates that the person has a high degree of catastrophizing pain.
Experimental (Skin cooling) Pain (Visual Analogue Pain Scale) | 4 week
  The visual analog pain scale will be used to measure pain in hemodialysis patients. The scale consists of a horizontal line 10 cm tall. A VAS score of 0, consisting of numerical values sorted on a horizontal line, indicates that there is no pain at all, while a score of 10 indicates the most severe pain. A pain rating of 0 on a scale with a rating between 0 and 10 in patients means that there is no pain, a pain rating of 1 to 3 Decrees mild pain, 4 to 6 moderate pain and a pain rating of 7 or higher Decrees severe pain.
Experimental (The valsalva maneuver group)The pain catastrophizing scale | 4 week
  This scale, developed by Sullivan et al. (1995), serves to measure the exaggerated negative mental reaction of individuals to an existing or predicted painful experience; to what extent they catastrophize the pain in the form of self-information.The reliability and validity of the Turkish version of the scale, which was shown by Uğurlu and others (2017), consists of 13 items. Each item is scored as none at all=0, mild degree=1, moderate degree=2, major degree=3 and always=4. A high total score indicates that the person has a high degree of catastrophizing pain
Experimental (The valsalva maneuver group) Pain (Visual Analogue Pain Scale) | 4 week
  The visual analog pain scale will be used to measure pain in hemodialysis patients. The scale consists of a horizontal line 10 cm tall. A VAS score of 0, consisting of numerical values sorted on a horizontal line, indicates that there is no pain at all, while a score of 10 indicates the most severe pain. A pain rating of 0 on a scale with a rating between 0 and 10 in patients means that there is no pain, a pain rating of 1 to 3 Decrees mild pain, 4 to 6 moderate pain and a pain rating of 7 or higher Decrees severe pain.
Experimental group (Antistress ball group) The Pain Catastrophization Scale | 4 week
  This scale, developed by Sullivan et al. (1995), serves to measure the exaggerated negative mental reaction of individuals to an existing or predicted painful experience; to what extent they catastrophize the pain in the form of self-information . The reliability and validity of the Turkish version of the scale, which was shown by Uğurlu and others (2017), consists of 13 items. Each item is scored as none at all=0, mild degree=1, moderate degree=2, major degree=3 and always=4. A high total score indicates that the person has a high degree of catastrophizing pain.
Experimental (Antistress ball group) Pain (Visual Analogue Pain Scale) | 4 week
  The visual analog pain scale will be used to measure pain in hemodialysis patients. The scale consists of a horizontal line 10 cm tall. A VAS score of 0, consisting of numerical values sorted on a horizontal line, indicates that there is no pain at all, while a score of 10 indicates the most severe pain. A pain rating of 0 on a scale with a rating between 0 and 10 in patients means that there is no pain, a pain rating of 1 to 3 Decrees mild pain, 4 to 6 moderate pain and a pain rating of 7 or higher Decrees severe pain.
Control group The Pain Catastrophization Scale | 4 week
  This scale, developed by Sullivan et al. (1995), serves to measure the exaggerated negative mental reaction of individuals to an existing or predicted painful experience; to what extent they catastrophize the pain in the form of self-information . The reliability and validity of the Turkish version of the scale, which was shown by Uğurlu and others (2017), consists of 13 items. Each item is scored as none at all=0, mild degree=1, moderate degree=2, major degree=3 and always=4. A high total score indicates that the person has a high degree of catastrophizing pain.
Control Group Pain (Visual Analogue Pain Scale) | 4 week
  The visual analog pain scale will be used to measure pain in hemodialysis patients. The scale consists of a horizontal line 10 cm tall. A VAS score of 0, consisting of numerical values sorted on a horizontal line, indicates that there is no pain at all, while a score of 10 indicates the most severe pain. A pain rating of 0 on a scale with a rating between 0 and 10 in patients means that there is no pain, a pain rating of 1 to 3 Decrees mild pain, 4 to 6 moderate pain and a pain rating of 7 or higher Decrees severe pain.

SECONDARY OUTCOMES:
Experimental(Skin cooling) Pain (Visual Analogue Pain Scale) | 8 week
  The visual analog pain scale will be used to measure pain in hemodialysis patients. The scale consists of a horizontal line 10 cm tall. A VAS score of 0, consisting of numerical values sorted on a horizontal line, indicates that there is no pain at all, while a score of 10 indicates the most severe pain. A pain rating of 0 on a scale with a rating between 0 and 10 in patients means that there is no pain, a pain rating of 1 to 3 Decrees mild pain, 4 to 6 moderate pain and a pain rating of 7 or higher Decrees severe pain.
Experimental (Skin cooling) The Pain Catastrophization Scale | 8 week
  This scale, developed by Sullivan et al. (1995), serves to measure the exaggerated negative mental reaction of individuals to an existing or predicted painful experience; to what extent they catastrophize the pain in the form of self-information. The reliability and validity of the Turkish version of the scale, which was shown by Uğurlu and others (2017), consists of 13 items. Each item is scored as none at all=0, mild degree=1, moderate degree=2, major degree=3 and always=4. A high total score indicates that the person has a high degree of catastrophizing pain
Experimental group (Valsalva Maneuver Group) Visual Analog Pain Scale | 8 week
  The visual analog pain scale will be used to measure pain in hemodialysis patients. The scale consists of a horizontal line 10 cm tall. A VAS score of 0, consisting of numerical values sorted on a horizontal line, indicates that there is no pain at all, while a score of 10 indicates the most severe pain. A pain rating of 0 on a scale with a rating of 0 to 10 in patients means that there is no pain, a pain rating of 1 to 3 means mild pain, 4 to 6 moderate pain, and a pain rating of 7 or higher means severe pain.
Experimental (The valsalva maneuver group) The Pain Catastrophization Scale | 8 week
  This scale, developed by Sullivan et al. (1995), serves to measure the exaggerated negative mental reaction of individuals to an existing or predicted painful experience; to what extent they catastrophize the pain in the form of self-information. The reliability and validity of the Turkish version of the scale, which was shown by Uğurlu and others (2017), consists of 13 items. Each item is scored as none at all=0, mild degree=1, moderate degree=2, major degree=3 and always=4. A high total score indicates that the person has a high degree of catastrophizing pain
Experimental(Antistress ball group) Pain (Visual Analogue Pain Scale) | 8 week
  The visual analog pain scale will be used to measure pain in hemodialysis patients. The scale consists of a horizontal line 10 cm tall. A VAS score of 0, consisting of numerical values sorted on a horizontal line, indicates that there is no pain at all, while a score of 10 indicates the most severe pain. A pain rating of 0 on a scale with a rating between 0 and 10 in patients means that there is no pain, a pain rating of 1 to 3 Decrees mild pain, 4 to 6 moderate pain and a pain rating of 7 or higher Decrees severe pain.
Experimental (Antistress ball group) The Pain Catastrophization Scale | 8 week
  This scale, developed by Sullivan et al. (1995), serves to measure the exaggerated negative mental reaction of individuals to an existing or predicted painful experience; to what extent they catastrophize the pain in the form of self-information. The reliability and validity of the Turkish version of the scale, which was shown by Uğurlu and others (2017), consists of 13 items. Each item is scored as none at all=0, mild degree=1, moderate degree=2, major degree=3 and always=4. A high total score indicates that the person has a high degree of catastrophizing pain
Control Group Pain (Visual Analogue Pain Scale) | 8 week
  The visual analog pain scale will be used to measure pain in hemodialysis patients. The scale consists of a horizontal line 10 cm tall. A VAS score of 0, consisting of numerical values sorted on a horizontal line, indicates that there is no pain at all, while a score of 10 indicates the most severe pain. A pain rating of 0 on a scale with a rating between 0 and 10 in patients means that there is no pain, a pain rating of 1 to 3 Decrees mild pain, 4 to 6 moderate pain and a pain rating of 7 or higher Decrees severe pain.
Control group The Pain Catastrophization Scale | 8 week
  This scale, developed by Sullivan et al. (1995), serves to measure the exaggerated negative mental reaction of individuals to an existing or predicted painful experience; to what extent they catastrophize the pain in the form of self-information. The reliability and validity of the Turkish version of the scale, which was shown by Uğurlu and others (2017), consists of 13 items. Each item is scored as none at all=0, mild degree=1, moderate degree=2, major degree=3 and always=4. A high total score indicates that the person has a high degree of catastrophizing pain

CONTACTS AND LOCATIONS:
Overall Officials: AYNUR CIN, DR, Principal Investigator — Gümüşhane Universıty
Locations (1):
- Kelkit State Hospital, Kelkit, Gümüşhane Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Study Protocol
Supporting Information: Study Protocol
Time Frame: 01.10.2024-31.12.2024
Access Criteria: It can be received by e-mail with the permission of the researcher.
URL: https://giris.tubitak.gov.tr/kullaniciadiilegiris.htm